CLINICAL TRIAL: NCT07203183
Title: A Prospective Study for the Collection of Whole Blood Samples to Support the Development and Validation of In Vitro Diagnostic Tests for Dengue
Brief Title: Dengue - Sample Collection Study Pakistan
Status: Not yet recruiting | Type: Observational
Sponsor: Abbott Rapid Dx (Industry)
Collaborators: Aga Khan University (Other); National University of Medical Sciences, Pakistan (Other)
Responsible Party: Sponsor
Other Study IDs: SDRD-K-029-P
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Dengue
Keywords: dengue; sample collection; serum; plasma; blood
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, no human genetic testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dengue positives
- dengue negatives

SUMMARY:
The objective of this study is to collect well-characterized serum and plasma specimens from confirmed dengue positive and dengue negative subjects to support dengue diagnostic products development.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12-years-old
* Individuals suspected or confirmed for active dengue, with dengue-consistent symptoms onset up to and including 10 days before enrolment in this trial.

Exclusion Criteria:

* Subject has been vaccinated for dengue.
* Subject participates in an investigative drug, vaccine or medical device clinical study
* Participant is deemed unfit for the study by the Investigator
* Participant is unwilling or unable to provide informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with symptoms suggestive of active dengue or a recent diagnosis of dengue seeking clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
sample collection only, no specific outcome needed | 5 months